CLINICAL TRIAL: NCT06157242
Title: A Phase 1, Open-label, Single-dose Study to Determine the Safety and Pharmacokinetics of ORAvance (Ceftibuten/Xeruborbactam Oral Prodrug [QPX7831]) in Participants With Renal Impairment
Brief Title: PK & Safety Study of Xeruborbactam Oral Prodrug Combined With Ceftibuten in Participants With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Qpex Biopharma, Inc. (Industry)
Collaborators: Shionogi Inc. (Industry); Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Qpex-103
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Bacterial Infections
Keywords: beta-lactamase inhibitor
MeSH Terms: conditions — Bacterial Infections | interventions — Ceftibuten

STUDY DESIGN:
Intervention Model Description: Open-label, single dose design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label, Single Dose Combination of Ceftibuten & Xeruborbactam oral prodrug (Experimental): 24 pts will be enrolled with varying degrees of RI as well as 8 participants with normal renal function (NRF). 8 participants will be enrolled in each group (G) based on estimated glomerular function rate (eGFR) at screening:
  * G1: Mild RI (eGFR 60 to 90 mL/min/1.73m2 calculated using the Chronic Kidney Disease Epidemiology Collaboration equation [CKP-EPI]) adjusted for the participant's body surface [BSA])
  * G2: Moderate RI (eGFR 30 to < 60 mL/min/1.73m2 calculated using the CKD-EPI equation adjusted for the participant's BSA)
  * G3: Severe RI (eGFR < 30 mL/min/1.73m2 calculated using the CKD-EPI equation) not receiving dialysis therapy
  * G4: Healthy participants with NRF matched to patients in Groups 1, 2 and 3 based on age, gender and BMI All pts will receive a single dose of ceftibuten & QPX7831 on Day 1. Pts will remain in the clinic until completion of the post-dose procedures on Day 8. Participants will be contacted by phone between Days 10-12 for follow-up.
  Interventions: Drug: Xeruborbactam Oral Prodrug; Drug: Ceftibuten

INTERVENTIONS:
Drug: Xeruborbactam Oral Prodrug — Experimental
  Other Names: QPX7831
Drug: Ceftibuten — Experimental

SUMMARY:
A Phase 1, open-label, single-dose study to determine the safety and pharmacokinetics of ORAvance (ceftibuten/xeruborbactam oral prodrug [QPX7831]) in participants with renal impairment

DETAILED DESCRIPTION:
Qpex Biopharma, Inc. is developing an oral dosage form that delivers Xeruborbactam, a new boron-based beta-lactamase inhibitor with activity against both serine and metallo-beta-lactamases, for oral treatment in combination with a beta-lactam antibiotic.

Ceftibuten is a cephalosporin antibiotic approved in the US for acute exacerbations of chronic bronchitis, acute bacterial otitis media and pharyngitis/ tonsillitis.

This is a Phase 1 open-label, single-dose study to assess the safety, tolerability, and PK, of ceftibuten and xeruborbactam oral prodrug given in combination to participants with varying degrees of renal impairment as compared to participants with normal renal function.

Objectives:

The objectives of the study are:

1. To assess the PK of ceftibuten and xeruborbactam oral prodrug given in combination in participants with varying degrees of renal impairment.
2. To evaluate the safety and tolerability of ceftibuten and xeruborbactam oral prodrug given in combination in participants with varying degrees of renal impairment.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

1. Able to understand the study conduct and tasks required of the participants, sign the informed consent form and willing to cooperate with all tests and examinations required by the protocol.
2. Males and females at least 18 years of age, at the time of consent.
3. If male, agree to be sexually abstinent or to use 2 approved methods of contraception (refer to Inclusion Criterion #4) when engaging in sexual activity from study check-in through 930 days following the last administration of the study intervention, and to refrain from donating sperm during this same period of time. If the sexual partner is surgically sterile, contraception is not necessary.
4. Females of childbearing potential must either be sexually abstinent for 14 days prior to day 1 and remain so through 30 days following the last administration of the study intervention, OR have been using (or agree to use) 2 acceptable methods of birth control for the times specified:

   1. Intra-uterine device in place for at least 3 months prior to day 1 through 30 days following the final dosing of the study intervention
   2. Barrier method (condom or diaphragm) for at least 14 days prior to day 1 through 30 days following the final dosing of the study intervention
   3. Stable hormonal contraceptive for at least 3 months prior to day 1 through 30 days following final dosing of the study intervention
   4. Surgical sterilization (vasectomy) of partner at least 6 months prior to day 1
5. Females of non-childbearing potential must either be postmenopausal (defined as 12 months spontaneous amenorrhea) with a serum follicle stimulating hormone (FSH) level in the laboratory defined postmenopausal range or have undergone 1 of the following sterilization procedures detailed in the study protocol at least 6 months prior to day 1:

   1. Bilateral tubal ligation
   2. Hysterectomy
   3. Hysterectomy with unilateral or bilateral oophorectomy
   4. Bilateral oophorectomy
6. Have a BMI ≥ 18.5 kg/m2 and ≤ 45 kg/m2, inclusive.
7. Have sufficient peripheral vascular access, based on the site's assessment, for PK blood sample collection.
8. Have a semi-recumbent pulse rate ≥ 45 beats per minute (bpm) and ≤ 110 bpm during the vital sign assessment at the screening visit or day -1.
9. Willing to abstain from alcohol for 48 hours prior to dosing through discharge from the phase 1 unit on day 8.

   Participants With Renal Impairment:
10. Have an eGFR < 90 mL/min calculated using the CKD-EPI equation adjusted for the participant's BSA and will be calculated using the estimation equation recommended by the FDA. Specifically, group 1, mild renal impairment (eGFR 60 < 90 mL/min); group 2, moderate renal impairment (eGFR 30 to < 60 mL/min); and group 3, severe renal impairment (eGFR < 30 mL/min) not receiving dialysis therapy.
11. Have negative test results for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibody and anti-human immunodeficiency virus (HIV) antibody. Participants with renal impairment with a positive HCV antibody result will be included at the investigator's discretion if all liver enzyme parameters are within the normal range.

    Participants With Normal Renal Function:
12. Have an eGFR ≥ 90 mL/min calculated using the CKD-EPI equation adjusted for the participant's BSA.
13. Have negative test results for HBsAg, anti HCV antibody and anti-HIV antibody.
14. Meet matching criteria for age, BMI, and gender of pooled renally impaired as defined in the protocol.

Exclusion Criteria:

All Participants:

1. Have unstable or new medical conditions (eg, cardiovascular, respiratory, hepatic, renal, gastrointestinal, autoimmune, endocrine, or neurological disorders) which have occurred in the 3 months prior to the first dose of study intervention and which are capable of altering the absorption, distribution, metabolism, or elimination of drugs or, in the opinion of the investigator, constitute a risk factor to participating in the study and/or receiving study intervention.
2. Documented hypersensitivity reaction or anaphylaxis to any antibiotic including ceftibuten or other beta-lactam antibiotics (eg, cephalosporins, penicillins, carbapenems, or monobactams) or any excipients used in this formulation.
3. History of clinically significant seizures, head injury, or meningitis.
4. Current evidence or history of malignancy, except squamous cell carcinoma or basal cell carcinoma of the skin, in the 2 years prior to day -1 with no evidence of recurrence.
5. Females who are pregnant, lactating, or have a positive pregnancy test at the screening visit or day -1.
6. Previously received any dose of ORAvance (ceftibuten/xeruborbactam oral prodrug), xeruborbactam oral prodrug, xeruborbactam or prodrug alone.
7. Received any investigational drug within 30 days or 5 half-lives, whichever is longer, prior to day 1 of the current study.
8. Blood donation or significant blood loss (ie, > 500 mL) within 56 days prior to day 1.
9. Plasma or platelet donation within 14 days prior to day -1.
10. Any acute illness requiring antibiotic drug therapy within 30 days prior to day 1 or a febrile illness within 7 days prior to day 1.
11. Vigorous exercise from 48 hours prior to day -1 until the day of discharge from the study.
12. Positive drug test at the screening visit or day -1 unless results can be explained by a prescription medication and/or recent history (ie, within 6 months prior to day -1) of abuse of prescription or illicit drugs as detailed in the study protocol.
13. Positive alcohol test at the screening visit or day -1 and/or recent history (ie, within 6 months prior to day -1) of excessive alcohol intake as defined in the study protocol.

    Excessive intake of alcohol, defined as an average weekly intake of > 14 standard drinks, (standard drink is the equivalent to 120 ml of wine (approximately 12% abv), 350 ml of regular beer (approximately 5% abv), or 45 ml of spirits (40% abv).
14. Concurrent use of medications known to affect the elimination of serum creatinine and competitors of renal tubular secretion within 30 days prior to the first dose of study intervention or anticipated need for these therapies through the last PK sample.
15. Employees of the investigative site involved in this study.
16. Unable or unwilling to adhere to the study-specified procedures and restrictions.
17. QTcF interval > 500 msec, previous history or family history of prolonged QT syndrome at screening or day -1.
18. Use of products containing caffeine, xanthine, or ephedrine within 24 hours before dosing; the use of alcohol 48 hours prior to dosing; or antacids including calcium carbonate, H2 receptor blockers, and proton pump inhibitors are prohibited 7 days prior to day 1 until the end of the study, including both over-the-counter (OTC) and prescription drugs in these categories.
19. Have any clinically significant abnormalities in laboratory values at screening or check-in (day -1), defined in the study protocol.
20. Liver function abnormalities at screening or check-in (day -1) (defined by an elevation in total bilirubin, aspartate aminotransferase (AST), or alanine transaminase (ALT), > upper limit of normal range for participants based on age and sex).

    Participants With Renal Impairment:
21. Abnormal and clinically significant findings on physical examination, medical history, serum chemistry, hematology, or urinalysis per investigator discretion. Participants in the renal impairment group will have consideration for the degree of renal impairment and presence of comorbidities.
22. Have a semi-recumbent systolic BP > 180 or < 90 mm Hg or have a semi-recumbent diastolic BP > 110 or < 50 mm Hg at the screening visit or day -1.

    Participants With Normal Renal Function:
23. Abnormal and clinically significant findings on physical examination, medical history, serum chemistry, hematology, or urinalysis per investigator discretion.
24. Have a semi-recumbent systolic BP > 150 or < 90 mm Hg or have a semi-recumbent diastolic BP > 95 or < 50 mm Hg at the screening visit or day -1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-11-10 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent adverse events by subject and by group | 10 days
  Number of patients with Treatment-Emergent Adverse Events by subject, by group, severity and relationship to treatment
Number of patients with changes from baseline in safety parameters | 10 days
  Number of patients with changes in safety parameters before and after dosing by subject and group
Peak plasma Concentration measurements by subject and by group (Cmax) | 10 days
  Comparison will be performed between the groups for concentration measurements (Cmax). Mean graphical presentation of the data will be reported.
  Statistical analysis of exposure parameters will be performed.
Time concentration data measurements by subject and by group (Tmax) | 10 days
  Comparison will be performed between the groups for time concentration data measurements (Tmax)
Area under the plasma concentration versus time curve (AUC) between groups | 10 days
  Comparison will be performed between the groups for area under the plasma concentration versus time curve (AUC) Mean graphical presentation of the data will be reported. Statistical analysis of exposure parameters will be performed.
Urine Pharmacokinetic (PK) amount excreted by subject and by group | 10 days
  Urine Pharmacokinetic (PK) parameters such as amount excreted will be calculated from urinary excretion data
Urine Pharmacokinetic (PK) % dose excreted by subject and by group | 10 days
  Urine Pharmacokinetic (PK) parameters such as amount of % dose excreted will be calculated from urinary excretion data

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Loutit, MBChB, Study Director — Qpex Biopharma, Inc.
Locations (2):
- United States (2):
  - University of Miami Clinical Pharmacology, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No